CLINICAL TRIAL: NCT03348878
Title: Drug Compliance of Patients With Uncontrolled Hypertension Under Treatment: a Pilot Study (Descriptive, Prospective, Monocentric Cohort)
Brief Title: Descriptive Study of Drug Compliance in Uncontrolled Hypertensive Patients
Acronym: THERMO-HTA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: only 4 patients
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL17_0325
Record Dates: First submitted 2017-11-16; First posted 2017-11-21 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Uncontrolled Hypertension
Keywords: drug compliance; hypertension; anti-hypertensive agents
MeSH Terms: conditions — Medication Adherence; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohort of uncontrolled hypertensive patients (Other)
  Interventions: Other: assessment of drug compliance

INTERVENTIONS:
Other: assessment of drug compliance — assessment of drug compliance using electronic monitoring devices (2 months duration)

SUMMARY:
Therapeutic compliance is defined as the degree of coincidence between a person's behavior and prescribing advice given by his or her physician. According to the World Health Organization (WHO), "insufficient adherence is the main reason why patients do not get all the benefits they could expect from their medicines. It causes medical and psychosocial complications, diminishes the quality of life of patients, increases the likelihood of drug resistance, and waste of resources. " In the case of certain conditions such as high blood pressure (hypertension), poor adherence increases the risk of stroke, acute coronary syndrome, and heart failure.

In patients with uncontrolled hypertension under treatment, the issue of therapeutic non-compliance should always be considered before considering the dose (supplemental drug) of antihypertensive therapy.

For each patient participating in the study, medication adherence (for one of the antihypertensive treatments) will be assessed for 2 months using an electronic pill. The antihypertensive treatments considered for the study belong to the following classes: diuretics, beta-blockers, calcium-blockers, ACE (angiotensin-converting enzyme) inhibitors, sartans.

Main objective: care objective: to provide physicians and patients with assistance in case of ineffectiveness or therapeutic escape in a chronic disease such as hypertension, by assessing the compliance profile of each patient.

Secondary objectives: to carry out a quantitative typology of drug adherence in patients with unbalanced HTA under treatment.

ELIGIBILITY:
Inclusion Criteria:

* patient treated with diuretics and / or beta-blockers and / or calcium-blockers and / or ACE inhibitors and / or sartans
* Holter blood pressure total average of 24h greater than 135/85 mmHg or a daytime average greater than 140/90 mmHg or a nighttime average greater than 125/75 mmHg.
* informed consent given

Exclusion Criteria:

* Adults with severe hypertension (BP ≥ 180/110 mmHg) with or without organ failure requiring therapeutic adaptation
* Adults unable to comply with study procedures
* Patients who do not wish to receive generic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
individual pattern of drug compliance | 2 months of follow-up
  compliance measurement using electronic monitoring devices

SECONDARY OUTCOMES:
Percentage of Prescribed Dosing Days with Correct Intake | 2 months of follow-up
  The percentage of days with accurate dose intake is defined according to the reference: Vrijens B, Goetghebeur E. Comparing compliance patterns between randomized treatments. Control Clin Trials. 1997 Jun;18(3):187-203.
Percentage of Prescribed Dose Taken | 2 months of follow-up
  This measure, though often close to the previous one, focuses on the dose actually received and is defined according to the reference: Vrijens B, Goetghebeur E. Comparing compliance patterns between randomized treatments. Control Clin Trials. 1997 Jun;18(3):187-203.
Percentage of Drug Holidays | 2 months of follow-up
  We define a "drug holiday" as a period of one or more days without drug intake (that is, without MEMS (Medication Event Monitoring System) opening). The statistic counts the number of gaps among the prescribed days, ignoring the length of each individual gap, according to the reference: Vrijens B, Goetghebeur E. Comparing compliance patterns between randomized treatments. Control Clin Trials. 1997 Jun;18(3):187-203.
Time Variability in Drug Intake | 2 months of follow-up
  summary measures consider only the number of medication events each day, according to the reference: Vrijens B, Goetghebeur E. Comparing compliance patterns between randomized treatments. Control Clin Trials. 1997 Jun;18(3):187-203.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: No